CLINICAL TRIAL: NCT07034222
Title: A 12-month Single-arm Real-world Study to Determine the Safety and Efficacy of Lecanemab in Patients With Early Alzheimer's Disease
Brief Title: 12-Month Real-World Safety & Efficacy of Lecanemab in Early Alzheimer's Disease
Status: Active, not recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Ruijin Hospital (Other)
Responsible Party: Principal Investigator, WENYAN KANG, Professor and Chief Physician, Department of Neurology, Ruijin Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2025025
Record Dates: First submitted 2025-06-03; First posted 2025-06-24 (Actual); Last update posted 2025-06-24 (Actual); Status verified 2025-06

CONDITIONS: Alzheimer's Disease(AD)
MeSH Terms: conditions — Alzheimer Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Lecanemab treatment group (Experimental): receive 10 mg/kg of Leqembi once every two weeks. Dissolve Leqembi in normal saline and administer it intravenously over 60 minutes.
  Interventions: Drug: Administer Leqemi 10 mg/kg, every two weeks.

INTERVENTIONS:
Drug: Administer Leqemi 10 mg/kg, every two weeks. — Receive 10 mg/kg of Leqembi once every two weeks. Dissolve Leqembi in normal saline and administer it intravenously over 60 minutes. The infusion system must use a 0.2-μM terminal line filter for administration.

SUMMARY:
This is a 12-month, single-arm, real-world study designed to evaluate the efficacy and safety of lecanemab (10 mg/kg administered every two weeks) in patients with early Alzheimer's disease, including mild cognitive impairment (MCI) due to AD or mild AD dementia, confirmed by amyloid-positive Aβ-PET scans. The study will enroll 80 participants, with both retrospective and prospective data collection.

DETAILED DESCRIPTION:
The study enrolled participants with mild cognitive impairment due to AD or mild AD. All participants received biweekly intravenous infusions of lecanemab at a dose of 10 mg/kg. Safety data was collected, particularly for amyloid-related imaging abnormalities (ARIA). Effectiveness evaluations included cognitive tests, plasma biomarker analysis, and advanced neuroimaging.

ELIGIBILITY:
Inclusion Criteria:

* Meets the NIA-AA 2011 diagnostic criteria for:

Mild Cognitive Impairment due to Alzheimer's Disease (MCI-AD) or Mild Alzheimer's Disease Dementia.

-Confirmed Aβ pathology by: Aβ-PET scan or CSF Aβ42/Aβ40 ratio (results within 6 months prior to screening).

-Cognitive scales (within 3 months): Clinical Dementia Rating (CDR) global score 0.5-1 and/or Mini-Mental State Examination (MMSE) score 20-30.

* APOE genotype results available.
* MRI/SWI eligibility:
* No exclusionary findings (see Exclusion Criteria for details).
* Laboratory tests within normal ranges or deemed non-clinically significant by the investigator:

Routine tests: Liver/kidney function, CBC, urinalysis, fecal occult blood. Thyroid function: Free T3, free T4, TSH. Vitamin B12 (and methylmalonic acid [MMA], if available). Coagulation panel: PT/INR, aPTT (required). Negative for syphilis, HIV, or other infections that may affect cognition.

Exclusion Criteria:

- MRI/SWI exclusionary findings: 4 microhemorrhages (maximum diameter ≤10 mm). Any macrohemorrhage (>10 mm in diameter). Cortical superficial siderosis. Vasogenic edema. Evidence of brain contusion, encephalomalacia, vascular malformations, or infectious lesions.

Multiple lacunar infarcts/strokes in major vascular territories, severe small vessel disease, or severe white matter lesions (Fazekas grade ≥3).

Space-occupying lesions or brain tumors (except asymptomatic meningiomas/arachnoid cysts <1 cm).

Ages: 50 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2024-02-01 (Actual); Primary Completion 2026-01-01 (Estimated); Study Completion 2026-01-01 (Estimated)

PRIMARY OUTCOMES:
Change in Amyloid Burden as Assessed by Aβ-PET Standardized Uptake Value Ratio (SUVR) | Baseline, 6 months, 12 months
  Measurement:
  Unit of Measure: SUVR (unitless ratio) Reference Region: Cerebellar gray matter Range: Typically 1.0-3.0 in amyloid-positive subjects Direction: Lower values indicate greater amyloid clearance
Change in Amyloid Burden as Assessed by Centiloid Scale | Baseline, 6 months, 12 months
  Measurement:
  Unit of Measure: Centiloids (CL)
  Scale Range:
  0 CL: Young healthy controls 100 CL: Typical Alzheimer's dementia threshold Direction: Lower values indicate greater amyloid clearance

SECONDARY OUTCOMES:
Incidence of treatment-emergent adverse events (TEAEs) | 0-12 months (continuous monitoring)
  Safety evaluation including:
  All adverse events (AEs) Hematological and biochemical laboratory abnormalities Vital sign changes ECG abnormalities ARIA (amyloid-related imaging abnormalities) monitoring via brain MRI with specific protocols for ARIA-H (hemorrhage) and ARIA-E (edema) management
Change in Cognitive Function as Assessed by Clinical Dementia Rating Scale Sum of Boxes (CDR-SB) | Baseline, 3 months, 6 months, 12 months
  Scale Details:
  Score Range: 0 (best) to 18 (worst) Boxes Assessed:Memory，Orientation，Judgment & Problem Solving，Community Affairs，Home & Hobbies，Personal Care Scoring: Each domain rated 0 (none) to 3 (severe) Higher Score Indicates: Worse cognitive/functional impairment
Change in Cognitive Function as Assessed by Alzheimer's Disease Assessment Scale-Cognitive Subscale (ADAS-Cog14) | Baseline, 3 months, 6 months, 12 months
  Comprehensive neuropsychological test battery Scale range: 0 (best) to 90 (worst) Higher score indicates greater cognitive impairment
Change in Cognitive Function as Assessed by Mini-Mental State Examination (MMSE) | Baseline, 3 months, 6 months, 12 months
  Mini-Mental State Examination (MMSE) Scale range: 0 (worst) to 30 (best) Higher score indicates better cognitive function
Change in Neuropsychiatric Symptoms as Assessed by Neuropsychiatric Inventory (NPI) | Baseline, 3 months, 6 months, 12 months
  Scale Details:
  Total Score Range: 0 (best) to 144 (worst) Subscale Range (Frequency × Severity): 0-12 per domain Higher Score Indicates: Worse neuropsychiatric symptoms
  Domains Assessed:
  Delusions, hallucinations, agitation/aggression, depression/dysphoria, anxiety, elation/euphoria, apathy/indifference, disinhibition, irritability/lability, motor disturbance, nighttime behaviors, appetite/eating
Change in Functional Abilities as Assessed by the Alzheimer's Disease Cooperative Study-Activities of Daily Living for Mild Cognitive Impairment (ADCS MCI-ADL) | Baseline, 3 months, 6 months, 12 months
  Scale Details:
  Score Range: 0 (worst) to 53 (best) Higher Scores Indicate: Better daily functioning (less impairment)
  Assessed Domains:
  Basic ADLs (e.g., eating, dressing) Instrumental ADLs (e.g., shopping, managing finances)
Change in Caregiver Burden as Assessed by the Zarit Burden Interview (ZBI) | Baseline, 3 months, 6 months, 12 months
  Scale Details:
  Score Range: 0 (no burden) to 88 (severe burden) Higher Scores Indicate: Worse caregiver distress
  Interpretation:
  0-20: Little to no burden 21-40: Mild to moderate burden 41-60: Moderate to severe burden 61-88: Severe burden

OTHER OUTCOMES:
Change in Plasma Aβ42/40 Ratio | Baseline, 3 months, 6 months, 12 months
  Technology: Single Molecule Array (Simoa™, Quanterix) digital immunoassay
Change in Plasma Phosphorylated Tau (p-tau181) | Baseline, 6 months, 12 months
  Single Molecule Array (Simoa™, Quanterix) digital immunoassay
Change in Plasma Neurofilament Light (NfL) | Baseline, 3 months, 6 months, 12 months
  Single Molecule Array (Simoa™, Quanterix) digital immunoassay
Change in Plasma Glial Fibrillary Acidic Protein (GFAP) | Baseline, 3 months, 6 months, 12 months
  Single Molecule Array (Simoa™, Quanterix) digital immunoassay

CONTACTS AND LOCATIONS:
Locations (1):
- Ruijin Hospital, Shanghai Jiao Tong University School of Medicine, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Kang W, Gao C, Li X, Wang X, Zhong H, Wei Q, Tang Y, Huang P, Shen R, Chen L, Zhang J, Fang R, Wei W, Zhang F, Zhou G, Yuan W, Chen X, Yang Z, Wu Y, Xu W, Zhu S, Zhang L, He N, Fang W, Zhang M, Zhang Y, Ju H, Bai Y, Liu J. Safety and effectiveness of lecanemab in Chinese patients with early Alzheimer's disease: Evidence from a multidimensional real-world study. Chin Med J (Engl). 2025 Nov 20;138(22):2907-2916. doi: 10.1097/CM9.0000000000003888. Epub 2025 Oct 27. PMID 41069006